CLINICAL TRIAL: NCT04047277
Title: Clinical Outcomes of Cognitive Behavioral Therapy for Nightmares in Children
Brief Title: Cognitive Behavioral Therapy for Nightmares in Children
Acronym: CBT-NC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: University of Tulsa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB9653
Record Dates: First submitted 2019-06-05; First posted 2019-08-06 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Nightmare
Keywords: Nightmares; Children; Trauma; CBT; Exposure; Relaxation; Rescripting; Cognitive; Behavioral; Therapy
MeSH Terms: conditions — Wounds and Injuries; Behavior | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Blinded randomization into 2 groups: Treatment & Waitlist Control. Treatment group receives treatment right away. Waitlist group receives treatment after 6 week wait.
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Right-Away (Experimental): Cognitive Behavioral Therapy using exposure, relaxztion, and rescripting - Child utilizes behavioral and cognitive therapy techniques of exposure therapy and cognitive restructuring.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Waitlist Control (No Intervention): Waitlist control group will complete pre and post assessments at beginning and end of wait period.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The manualized CBT protocol is five sessions that teach sleep hygiene, relaxation strategies, and addresses nightmares therapeutically through exposure and rescripting.
  Arms: Treatment Right-Away

SUMMARY:
Up to 50% of children experience nightmares annually. Nightmares interfere with sleep quality and quantity resulting in sleep deficiency, and are associated with negative mental health consequences. Previous research has shown efficacy of manualized CBT treatment for reducing trauma related nightmares in adults, and preliminary evidence has shown efficacy in children. This study is the first randomized clinical trial to evaluate the effectiveness of the treatment for idiopathic, as well as trauma related nightmares in children. The treatment in a manualized CBT protocol (5 sessions) that teaches sleep hygiene, relaxation strategies, and addresses nightmares therapeutically through exposure and rescripting.

ELIGIBILITY:
Inclusion Criteria:

* Children must have a history of nightmares occurring approximately once or more per week over a minimum of one month.
* Children must have verbal comprehension of at least age 5 (determined by PPVT), and be fluent in English.
* If taking psychotropic medications, must be stable for one month.
* Children must have a parent or legal guardian who is able to participate in treatment assignments and be able to read and speak English.

Exclusion Criteria:

* Under age 5 or over age 17.
* No nightmares (or less than averaging one per week)
* Apparent psychosis
* Pervasive developmental disorder or mental retardation
* Not able to read and speak English.
* Sleep apnea

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change on the Child Adolescent Trauma Screen (CATS) - Child Version | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The CATS screens for child trauma history and PTSD symptoms in youth ages 7-17; 15 YES/NO questions; 1 open-ended question
Change on the Trauma Related Nightmare Survey (TRNS-C) - Child Version | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The TRNS-C is a 14 item self report measure that assesses current sleep quality, frequency, severity, and duration of nightmares, as well as cognitions, emotions, and behaviors related to nightmares in children.
Change on the Nightmare Distress Questionnaire (NDQ) | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The NDQ is a 13 item self report measure of nightmare related distress. Higher scores are significantly related to interest in therapy for nightmares.
Change on the Nightmare Locus of Control (NLOC) | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The N-LOC is an 6 item self report. This scale is collected as a child self report, and a caregiver report regarding child.
Change on the Pittsburgh Sleep Quality Index - Modified (PSQI) - Child Version | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The PSQI-M is a 10 item (with 2 items containing 23 sub items) self report measure of sleep quality and disturbance. It queries sleep quality and disturbances over the last month.
Change on the Children's Report of Sleep Patterns (CRSP) | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The CRSP is a 62 item self report measure of children's sleep patterns, sleep hygiene, and sleep disturbances for children eight to 12 years of age
Change on the Sleep Locus of Control (SLOC) | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The SLOC is an 6 item self report measure perceived contingencies between sleep behavior and events. This scale is collected as a child self report, and a caregiver report regarding child.
Change on the Epworth Sleepiness Scale (ESS) | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The ESS is an 8 item self report. The test is a list of eight situations in which one rates his/her tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. When the test is finished, response values are added up. The total score is based on a scale of 0 to 24. The scale estimates whether one is experiencing excessive sleepiness that possibly requires medical attention.
Change in reports on Sleep Journal | Participants complete this assessment at Pre-treatment (for 1 week), daily during the treatment phase, at Post treatment (for 1 week), at 3 month follow-up (for 1 week), and at 6 month follow-up (for 1 week).
  6 question self report that patient assesses daily from home.
Change on the Child Adolescent Trauma Screen (CATS) - Caregiver Report regarding child | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  The CATS screens for child trauma history and PTSD symptoms (information obtained from the caregiver, about the child).
Change on the Children's Sleep Habits - Caregiver Report regarding child | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  To examine sleep habits and possible difficulties with sleep in preschool and school-aged children
Adverse Childhood Experiences for CHILD - Caregiver Report regarding child | approximately 3 years.
  Assesses adverse experiences from infancy through early childhood
Change on the Sleep Disturbances Scale for Children - Caregiver Report regarding child | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  SDSC is a 26-item inventory rated on a 5 point Likert-type scale. The instrument's purpose is to categorize sleep disorders in children

SECONDARY OUTCOMES:
Change on the Parental Stress Scale | Participants will be assessed at Baseline (Week 0) through study completion, an average of 6 months.
  18 item self report scale used for the assessment of parental stress for both mothers and fathers and for parents of children with and without clinical problems. • 5 - Point scale; strongly disagree, disagree, undecided, agree, strongly agree. A low score signifies a low level of stress, and a high score to signifies a high level of stress.
Adverse Childhood Experiences for SELF - Caregiver Report regarding self | approximately 3 years.
  Assesses adverse experiences from infancy through early childhood

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Cromer, PhD, Principal Investigator — University of Tulsa; Tara R Buck, MD, Principal Investigator — University of Oklahoma School of Community Medicine
Locations (2):
- United States (2):
  - University of Tulsa, Tulsa, Oklahoma
  - University of Oklahoma School of Community Medicine, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No